CLINICAL TRIAL: NCT04772378
Title: An Intermediate Size Patient Population Expanded Access IND to Evaluate the Safety of Autologous HB-adMSCs for the Treatment of Patients With Parkinson's Disease.
Brief Title: Intermediate Size Patient Population Expanded Access IND for the Treatment of Patients With Parkinson's Disease.
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBPD05
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
Keywords: Mesenchymal Stem Cells; Parkinson's Disease; MSCs; Stem Cells; Neurodegenerative; Parkinson
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSCs — HB-adMSCs (Hope Biosciences autologous adipose-derived mesenchymal stem cells) is manufactured by Hope Biosciences, L.L.C., a biotechnology company headquartered in Sugar Land, Texas.

SUMMARY:
This Expanded Access IND is to evaluate the safety of multiple intravenous administrations of HB-adMSCs for treating Parkinson's disease in 10 patients between 76 and 95 y/o who do not qualify for other investigations.The dose to use for this expanded access is 200 million HB-adMSCs, administered through intravenous infusion only, with a treatment duration of 18 weeks. The program includes an up to 28 days screening period, an 18-week Treatment Period, and a 6-week Safety Follow-up Period.

DETAILED DESCRIPTION:
This expanded access program is designed to include adult male and female outpatients with Parkinson's disease with ages between 76 and 95 y/o.

-Screening During the Screening Visit, each patient who participates in the expanded access program must sign an informed consent form that the IRB has approved before any related procedures can be performed.

In addition to completing the informed consent process, the designated personnel are responsible for conducting the evaluations listed in the Schedule of Assessments. These evaluations include the following:

* Collection of vital signs, demographic information, and concomitant medications.
* Evaluation of the eligibility requirements for participation in the expanded access program.
* Weight and height measurements.
* Lab sample collection. (Comprehensive Metabolic Panel, Complete Blood Count & Coagulation Tests).
* Physical examination.
* Parkinson's disease assessments. (MDS-UPDRS, PDQ-39, PFS-16, PHQ-9, and VAS). Once these assessments have been performed and the results of laboratory tests have been obtained, the principal investigator must evaluate whether the screened patient is eligible to participate in the expanded access program. If a participant meets the eligibility requirements for participation in the expanded access program, infusion number 1 (the baseline visit) must be scheduled.

  * Infusions Every patient who qualifies for participation in the expanded access program will be invited to receive autologous HB-adMSCs infusions. The administration of investigational products will take place at the Hope Biosciences Stem Cell Research Foundation, where the delegated personnel will closely monitor patients' vital signs.

Following the Sponsor Standard Operating Procedures, Hope Biosciences autologous adipose- derived mesenchymal stem cells should be mixed and administered to each eligible patient. HB-adMSCs should only be administered intravenously and a vital sign monitoring of two hours post-drug exposure. Monitoring intervals of 0, 15, 30, 45, 60, 90, and 120 minutes.

Additional to the administration of the investigational product, the delegated personnel should complete the following assessments.

* Collection of vital signs, as well as updates on medical history and concomitant medications if needed.
* Weight measurement.
* Collection of laboratory samples at INF 1 and INF 5. (Comprehensive Metabolic Panel, Complete Blood Count& Coagulation Tests).
* Physical examination.
* Parkinson's disease assessments. (MDS-UPDRS, PDQ-39, PFS-16, PHQ-9, and VAS).
* Video documentation at INF 1 and INF 5 to evaluate the patient's gait, facial expression, and other symptoms associated with the disease.
* Determination of the incidence of AEs and SAEs. Immediately following the completion of each infusion, the patient should be assessed to ensure that the post-infusion discharge criteria have been met.

  * Follow Up A follow-up will be conducted during this visit. Delegated personnel will communicate with the patient to determine whether any adverse events or serious adverse events have occurred since the last visit. Also, during this visit, updates on medical history and concomitant medications must be recorded in the patient's chart if needed.
  * End of Expanded Access Program

Patients will be assessed by delegated personnel on the last visit of the expanded access program, which will take place at week 26. The following assessments will be performed:

* Collection of vital signs, as well as updates on medical history and concomitant medications if needed.
* Weight measurement.
* Collection of laboratory samples. (Comprehensive Metabolic Panel, Complete Blood Count& Coagulation Tests).
* Physical examination.
* Parkinson's disease assessments. (MDS-UPDRS, PDQ-39, PFS-16, PHQ-9, and VAS).
* Video documentation to evaluate the patient's gait, facial expression, and other symptoms associated with the disease.
* Determination of the incidence of AEs and SAEs.

ELIGIBILITY:
Inclusion Criteria

A participant will be eligible for inclusion in this expanded access program only if all the following criteria apply:

1. Patients aged 76-95 years old (male and female).
2. Patients must have had a Parkinson's disease diagnosis for a minimum of six months before 1st infusion.
3. Patients must have previously banked their mesenchymal stem cells with Hope Biosciences.
4. Patients should be able to read, understand, and provide voluntarily written consent.
5. Patients able and willing to comply with the requirements of this expanded access program.

Exclusion Criteria

A participant will not be eligible for inclusion in this expanded access program if any of the following criteria apply:

1. Patients with advanced Parkinson's disease. Advanced PD is defined as a significant disability, wheelchair-bound or bedridden.
2. Any malignancy or clinical evidence that supports the presence of a malignant process in a patient is being investigated. Malignancy is defined as any form of cancer that had occurred in the previous five years before the first infusion and may require surgery, chemotherapy, or radiation.
3. Patients with medical history of uncontrolled high blood pressure defined as a deficient standard of care treatment and/or blood pressure > 140/90 mm/Hg during screening visit.
4. Patients with the following concomitant or past medical history:

   * Heart Failure - New York Heart Association (NYHA) Class III/IV.
   * Heart Attack (in the past six months before 1st infusion).
   * Stroke (in the past six months before 1st infusion).
   * Hepatitis B or C.
   * Human immunodeficiency virus (HIV) infection.
5. Any of the following abnormal lab findings during screening will disqualify a patient from this expanded access program:

   * Hemoglobin (Hgb) <10 G/DL or >18 G/DL
   * Hematocrit (HCT) <30% or >54 %
   * Platelet count < 80 K/UL and or > 450 K/UL.
   * White blood cell count WBC < 3.0 K/UL and > 12.0 K/UL.
   * Alanine aminotransferase (ALT) of > 75 IU/L
   * Aspartate aminotransferase (AST) of > 75 IU/L
   * eGFR < 59 mL/min/1.73
   * Pre-prandial glucose > 130 MG/DL
   * Post-prandial glucose > 200 MG/DL
6. Patients who have received any stem cell treatment in the past six months before 1st infusion other than stem cells produced by Hope Biosciences.
7. Patients who are unlikely to complete the visits or adhere to the procedures.
8. The patient has previously been diagnosed with a psychiatric disorder, which is currently uncontrolled.
9. Patients with a history of addiction or dependency or currently abusing or using substances.
10. Patients with any form of kidney dialysis will be excluded from participation in the investigation.
11. Patients who have received an experimental drug in the past 12 months before the first dose of the investigational product. (Except for COVID-19 vaccinations).
12. Patients who the Investigator determines to be unsuitable for participation for other reasons, such as, but not limited to deep vein thrombosis (DVT), pulmonary embolus, cardiac arrhythmia, or those who have a prothrombotic condition, or who require persistent oxygen supplementation.
13. Patients who have recently undergone major surgery (in the past six months before 1st infusion). Some examples of major surgeries include, but are not limited to, the following: heart surgeries, aortic aneurysm bypass, organ transplant, intracranial surgery, spinal laminectomy or fusion, amputation, resection of the lung, resection of esophagus, resection of a mediastinal mass, resection of bladder or prostate tumor and resection of kidney or ureter.

Ages: 76 Years to 95 Years | Sex: All
Age Groups: Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States

REFERENCES:
- See also: Hope Biosciences Stem Cell Research Foundation — https://www.hopebio.org/